CLINICAL TRIAL: NCT05524870
Title: Movement With Mobilization Technic Plus Exercising Versus Exercising Alone for Central Sensitization in Patients With Subacromial Pain: a Sham-controlled Randomized Clinical Trial
Brief Title: The Effect of Manual Therapy on Central Sensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, Director, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107/82
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Subacromial Pain Syndrome; Central Sensitisation
Keywords: Manual therapy; Shoulder pain; Mobilization
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobilization (Experimental): Mobilization with movement plus exercise.
  Interventions: Other: Mobilization
- Sham mobilization (Placebo Comparator): Sham mobilization with movement plus exercise
  Interventions: Other: Mobilization
- Control (Active Comparator): Exercise alone
  Interventions: Other: Mobilization

INTERVENTIONS:
Other: Mobilization — Movement with mobilization plus exercise

SUMMARY:
Subacromial pain syndrome (SIS) is a common cause of shoulder pain, estimated to be the cause for up to half of incident cases. Typically, pain is generated with elevation of the arm above the head though it can occur with rest in patients with SIS.There is evidence of central sensitization in those who experience chronic shoulder pain from SIS. Central sensitization is an augmentation of the nociceptive pathways of the central nervous system that is characterized by local and generalized lowered pain thresholds and an exaggerated pain response to painful and non painful stimulation.Mobilization with movement (MWM) technic is a kind of manual therapy and it is often used by clinicians for the treatment of musculoskeletal diseases. Usually manual therapy is used for its peripheral effects, however it also produces central analgesic effects activating descending anti-nociceptive pathways for a short period of time (30 - 35 mins.). Some speculate that repeated sessions of manual therapy may result in a long term activation of descending anti-nociceptive pathways. However, there is no evidence of this mechanism available yet. Therefore, the aim of this study is to investigate the effect of MWM on central sensitization (primary aim) and shoulder functions (secondary aim) in patients with SIS.

ELIGIBILITY:
Inclusion Criteria:

* To have confirmed unilateral subacromial pain (positive testing at Neer Impingement and Hawkins-Kennedy tests),
* To have <40 score in central sensitization inventory.

Exclusion Criteria:

* To have bilateral subacromial pain,
* To have any pathology (except subacromial pain) that give rise to central sensitization (This pathologies are summarized in central sensitization inventory - part B)
* To have severe osteoarthritis or subluxation in shoulder joint,
* To have adhesive capsulitis,
* Being treated with physiotherapy for this disorder at least one month before the start of the study.
* To have severe cervical or lumbar radiculopathy,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory | Baseline, 3 weeks: change from baseline central sensitization at 3 weeks, 3 months: change from central sensitization at 3 months.
  The central sensitization inventory (CSI), a patient reported outcome measure, is a reliable and valid comprehensive screening instrument for identification of central sensitization. The CSI inventory comprises of two sections - Part A and Part B. Part A consisted of 25-item self-report questionnaire with each item assessed on a 5-point Likert scale (0=never and 4=always), with total scores ranging from 0-100. Part B evaluates health-related symptoms that are common to central sensitization syndromes.Higher scores indicate more severe central sensitization. A CSI cut-off score of 40 exhibited good sensitivity in identifying central sensitization.
Pressure-Pain Threshold-Algometer | Baseline, 3 weeks: change from baseline pressure pain threshold at 3 weeks, 3 months: change from pressure pain threshold at 3 months.
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure where a sense of pressure first changes to pain. A mechanical pressure algometer is used in this study to assess PPT. This device consists of a round rubber disk (area,1 cm2 ) attached to a pressure (force) gauge. The gauge displays values in kilograms. Because the surface of the rubber tip is 1 cm2, the readings are expressed in kilograms per square centimeter. The range of the algometer is 0 to 10 kg with 0.1-kg divisions. Higher scores indicate high PPT.

SECONDARY OUTCOMES:
Quick Disabilities of the Shoulder, Arm and Hand Questionnaire | Baseline, 3 weeks: change from baseline shoulder functions at 3 weeks, 3 months: change from shoulder functions at 3 months.
  The Quick Disabilities of the Shoulder, Arm and Hand Questionnaire assesses physical functioning and symptoms of the upper limb, yielding a result between 0 and 100% (0% being the best and 100% being the worst outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)